CLINICAL TRIAL: NCT06983197
Title: Iatrogena bristtillstånd Hos intensivvårdade Patienter Under långvarig Behandling Med Kontinuerlig Dialys
Brief Title: Iatrogenic Deficiencies in ICU Patients With Prolonged Continuous Renal Replacement Therapy
Acronym: IBRIST
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Grip, MD, PhD, Karolinska University Hospital
Other Study IDs: 2024-07642-01
Record Dates: First submitted 2025-04-30; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma is sampled and stored in -80 degress C before analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CRRT patients: Patients, all ages, that receive CRRT for at least five days.
  Interventions: Diagnostic Test: blood test
- Non-CRRT patient: Adult patients, >17 yo, treated in the ICU for 10-15 days without renal replacement therapy
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — Blood samples are drawn every 3-5 days in the RRT group but only once in the control group

SUMMARY:
ICU patients are recruited after at least 5 days treatment with continuous renal replacement therapy. Blood samples are drawn at time of recruitment and then every 3-5 days until ceseation of renal replacement therapy.

Samples will be analyzed for concentrations of trace elements, vitamins and amino acids.

10 adult ICU patients treated for two weeks without renal replacement therapy will be sampled at one time point to serve as controls.

ELIGIBILITY:
Inclusion Criteria CRRT group:

* CRRT more than 5 days

Exclusion Criteria:

* N/A

Inclusion criteria non-CRRT group

- ICU care 10-15 days without any dialysis treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient of all ages treated with CRRT
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of trace element | From enrollment to the end of treatment at 4 weeks
  Measurments of trace elements and vitamins as compared to established reference values as well as non-CRRT controls

SECONDARY OUTCOMES:
Amino acids | From enrollment to the end of treatment at 4 weeks
  Concentration of amino acids in plasma
Vitamins | At all measuring points
  Water soluble vitamins, concentration in plasma. Compared to non-crrt controls and established references

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grip, MD, PhD, Principal Investigator — Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: No
Data will be availible upon reasonable request but the small sample size number and specificity of medical conditions makes blinding to challenging for public release